CLINICAL TRIAL: NCT04991259
Title: To Evaluate the Safety and Efficacy of Preemptive Administration of Continuous Renal Replacement Therapy in Patients With Acute Liver Failure With Cerebral Edema -A Prospective Randomized Controlled Trial
Brief Title: To Evaluate the Safety and Efficacy of Preemptive Administration of Continuous Renal Replacement Therapy in Patients With Acute Liver Failure With Cerebral Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-05
Record Dates: First submitted 2021-06-25; First posted 2021-08-05 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-06

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive CRRT (Experimental): In patients randomized to early CRRT, CRRT would be initiated within 12 hours of randomization.
  Interventions: Procedure: Continuous Renal Replacement Therapy (CRRT)
- Standard Medical Treatment (Active Comparator): In patients randomized to SMT group, CRRT would be initiated as per the existing standard protocol.
  1. in patients with worsening hyperammonemia despite two sessions of plasma-exchange
  2. patients meeting renal indications (hyperkalemia, volume overload, oliguria or metabolic acidosis etc).
  Interventions: Procedure: Continuous Renal Replacement Therapy (CRRT); Other: Standard Medical Treatment

INTERVENTIONS:
Procedure: Continuous Renal Replacement Therapy (CRRT) — Continuous renal replacement therapy will be administered as continuous venovenous hemodiafiltration (CVVHDF) using Prisma and Prismaflex (Gambro) devices, with blood flows ranging from 150-180 mL/hr and target effluent rates of 20 - 25 mL/kg/hr. Anticoagulation was not used during dialysis. CRRT would be continued until resolution of cerebral edema and in decrease in ammonia levels below 150 ug/dl or in those who develop adverse effects of therapy.
Other: Standard Medical Treatment — In the L- ICU, patients will be managed by a multidisciplinary team. Intubation and ventilation will be undertaken for standard indications in addition to the development of grade 3 encephalopathy or evidence of cerebral edema on CT-scan. Fluid management will be done with crystalloids, with the use of colloids (5% albumin) in patients with severe hypoalbuminemia (serum albumin less than 2.5gm/dl). Norepinephrine will be the primary vasopressor used to target a mean arterial pressure of 65-70 mm of Hg. with adjunctive use of intravenous low dose hydrocortisone and vasopressin in patients not responsive to initial therapy.
  Arms: Standard Medical Treatment

SUMMARY:
In this prospective randomized controlled trial, investigator aim to evaluate the impact of early initiation of CRRT on outcomes in patients with acute liver failure with cerebral edema and hyperammonemia in improving cerebral edema and clinical outcomes. Investigator also aim to evaluate the effects of early initiation of CRRT on systemic hemodynamics (cardiac output and systemic vascular resistive index, extravascular lung water and lung permeability index), endothelial function and coagulation, microcirculation (as assessed by lactate clearance and central venous oxygen saturation), mitochondrial function. Patients with ALF who meet the inclusion and exclusion criteria.

Group 1: CRRT initiation within the first 12 hours Group 2: CRRT would be initiated i) In patients with worsening hyperammonemia despite two sessions of plasma-exchange ii) Patients meeting renal indications (hyperkalemia, volume overload, oliguria or metabolic acidosis etc)

DETAILED DESCRIPTION:
Hypothesis: Investigator hypothesize that preemptive administration of continuous renal replacement therapy would be synergistic to plasma-exchange in ameliorating the cytokine storm, cerebral edema and improve outcomes in patients with non-acetaminophen ALF with cerebral edema compared to late initiation.

Aim and Objective -

AIM:

Primary

1) 21-day transplant free survival with Prometheus Secondary

1. To compare the improvement effect in cerebral edema and hepatic encephalopathy in both groups
2. To study the safety of therapy (incidence of intradialytic hypotension, impairment of coagulation, hypothermia)
3. Duration of mechanical ventilation and ICU stay in both groups
4. Impact on arterial lactate
5. Improvement in SIRS
6. Effect on systemic hemodynamics and pulmonary function
7. Effect on endotoxin, DAMPS, pro-inflammatory cytokines, endothelial functions and coagulation

Methodology Study Protocol

All patients will be evaluated as follows:

* Clinical history and examination
* Etiology of acute event
* Severity assessment indices
* Complications if any Investigations Arterial blood gas analysis
* Hematology

  * CBC, Prothrombin time and INR
  * Peripheral smear, Retics
  * Thromboelastogram(ROTEM)
  * S.Fibrinogen level
* Biochemistry

  * Liver function testing
  * Kidney function test
  * Arterial ammonia levels
  * Serum lactate
  * CRP and procalcitonin
  * S.Ferritin and LDH
* Etiology of acute event:

  * Infectious etiology: IgM anti HAV, IgM anti HEV, IgM anti HBc ( If HBsAg +ve), IgM anti HDV ( If HBsAg +ve) , total antiHBc, anti HCV
  * Non Infectious etiology: Alcohol binging in last 4 weeks, hepatotoxic drugs, ANA (>1: 80), IgG
  * Non infectious etiology: Autoimmune markers, copper studies, iron studies, HOMA IR, FBS Imaging USG abdomen with Doppler for spleno-portal axis NCCT abdomen and brain Assessment of cerebral edema

    1. Optic nerve sheath diameter
    2. Transcranial doppler
    3. Electroechocardiogram

Study Population: 60 patients with ALF will be randomized to two groups in 1:1 ratio.

Study Design:

* A randomized controlled study.
* The study will be conducted on patients admitted to Department of Hepatology from May 2021 to March 2023 at ILBS, New Delhi
* Study group will comprise of patients with acute liver failure (ALF) with documented cerebral edema on CT-scan and arterial ammonia >150 ug/dl Study Period: May 2021 to March 2023 Sample Size calculation: Currently there are lack of studies investigating the timing of CRRT in patients with ALF therefore a minimum of 60 patients 30 in each group would be included in the current study.

The detailed cytokine profile, endotoxin assay, markers of endothelial dysfunction and bioenergetics would be performed in a subset of 10 patients in each group.

Intervention: Continuous renal replacement therapy

Monitoring and Assessment: Hourly till the patient is in the intensive care unit then every 7 days for 1 month

Statistical analysis

* All variables shall be expressed in median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables - Chi-Square or Fisher's test
* Survival analysis will be done using cox-proportional regression analysis
* Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.

Standard medical treatment: All patients will undergo plain CT-scan of the brain to screen for the presence and severity of cerebral edema in the emergency before being shifted to the L-ICU. In the L- ICU, patients will be managed by a multidisciplinary team. Intubation and ventilation will be undertaken for standard indications in addition to the development of grade 3 encephalopathy or evidence of cerebral edema on CT-scan. Ventilation will be managed by fentanyl and propofol along with the use of atracurium for paralysis wherever required. All patients will be monitored constantly for macro-hemodynamics, global tissue perfusion, and microcirculation. The macro-hemodynamic parameters included continuous monitoring of mean arterial pressure (MAP), heart rate and urine output per hour. The real-time monitoring of systemic vascular resistance (SVR), stroke volume variation (SVV), cardiac index (CI) and cardiac output (CO) will be done by a hemodynamic monitor (FloTrac™ system 4.0, Edwards Lifesciences, California, US) wherever feasible. Global tissue perfusion adequacy and indirect assessment of microcirculation will be done by measurement of arterial lactate. Fluid management will be done with crystalloids, with the use of colloids (5% albumin) in patients with severe hypoalbuminemia (serum albumin less than 2.5gm/dl). Norepinephrine will be the primary vasopressor used to target a mean arterial pressure of 65-70 mm of Hg. with adjunctive use of intravenous low dose hydrocortisone and vasopressin in patients not responsive to initial therapy.

Cerebral edema: The monitoring of cerebral edema will be performed measuring the optic nerve sheath diameter (ONSD) in both the eyes using a 7.5 MHz probe every 6-8 hours. Apart from this, routine monitoring of pupillary size and reactions, extensor posturing and plantar reflexes will be performed every 6-8 hrs. Transcranial doppler would be done every 6-8 hours. Patients will receive 3% hypertonic saline as a continuous infusion, initially started at 25ml /hr and titrated 6 hourly to between 5 and 20 mL per hour (maximum 100 ml/hour) to achieve serum sodium levels between 145-150 mmol/L. Intravenous 20% mannitol (1 g/kg IV bolus) over 20 to 30 minutes will be administered to those without renal failure. All patients will in addition receive intravenous N-acetylcysteine for 5 day.Routine electroencephalogram (EEG) will be done for all patients daily to screen for non-convulsive seizures which will be managed by intravenous levetiracetam. Assessment of coagulation will be performed by ROTEM at baseline and subsequently as required.

Protocol for standard-volume plasma-exchange

1. Standard-Volume Plasma Exchange: SVPE procedures will be performed using either Spectra Optia (SPO, Terumo BCT, Lakewood, CO, USA) continuous-flow centrifugal apheresis system or Haemonetics MCS+ (Braintree, MA, USA) intermittent flow centrifugal apheresis system via a double-lumen central venous dialysis catheter. All patients will receive plasma-exchange within first 6 hours of admission to the L-ICU along with a target volume of 1.5 to 2.0 plasma volumes per session. The replacement fluid used will be 90% FFP and 10% normal saline.PE will be performed on consecutive days until the desired response is achieved. [using investigator previously published protocol].
2. The number of sessions of SVPE in each patient will be decided based on the clinical response to SVPE. Dynamic assessment of the clinical parameters (signs of CE as assessed by pupillary size, reaction, and optic nerve-sheath diameter), INR, lactate and arterial ammonia will be performed at after each TPE. In patients with an improvement in INR, and signs of CE along with a reduction in ammonia at 6 hours which was sustained at 12 and 24 hours post-SVPE, subsequent sessions will be discontinued. PE will also be discontinued in patients who would show worsening in either clinical and/ or biochemical parameters. In patients who will develop adverse events, the PE procedure will be resumed or discontinued depending on the severity of adverse event and its resolution.

Randomization will be done by taking 1:1 ratio by computer-generated sealed envelopes by the clinical trial co-ordinator Group 1-Preemptive CRRT: In patients randomized to early CRRT, CRRT would be initiated within 12 hours of randomization.

Group 2: SMT - In patients randomized to SMT group, CRRT would be initiated as per the existing standard protocol.

in patients with worsening hyperammonemia despite two sessions of plasma-exchange patients meeting renal indications (hyperkalemia, volume overload, oliguria or metabolic acidosis etc).

The time to initiation of CRRT would be recorded in both groups after randomization.

Continuous renal replacement therapy will be administered as continuous venovenous hemodiafiltration (CVVHDF) using Prisma and Prismaflex (Gambro) devices, with blood flows ranging from 150-180 mL/hr and target effluent rates of 20 - 25 mL/kg/hr. Anticoagulation was not used during dialysis. CRRT would be continued until resolution of cerebral edema and in decrease in ammonia levels below 150 ug/dl or in those who develop adverse effects of therapy.

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute liver failure defined patients with jaundice which is complicated by encephalopathy and coagulopathy within 4 weeks of the onset of jaundice and without underlying chronic liver disease with documented cerebral edema on CT-scan and arterial ammonia >150 ug/dL.

Exclusion Criteria:

1. Age <18 or > 70 years
2. Hepatocellular Carcinoma
3. Active untreated Sepsis/DIC
4. Hemodynamic instability requiring high dose of vasopressors
5. Post-resection and malignancy related liver failure
6. Coma of non-hepatic origin
7. Patients with post renal obstructive AKI, AKI suspected due to glomerulonephritis, interstitial nephritis or vasculitis based on clinical history and urine analysis
8. Patients already meeting emergency criteria for immediate initiation of dialysis at the time of randomization (serum potassium>6 meq/lt, metabolic acidosis ph<7.12, acute pulmonary edema, severe volume overload with hypoxemia non-responsive to diuretic treatment)
9. Patients transferred from other hospitals who have already been on hemodialysis before their arrival in the intensive care unit
10. Extremely moribund patients with an expected life expectancy of less than 24 hours
11. Pregnancy related liver failure
12. Patients with significant renal dysfunction meeting absolute criteria for initiation of dialysis
13. Comorbidities associated with poor outcome (Extrahepatic neoplasia, severe cardiopulmonary disease defined by a New York Heart Association score >3, or oxygen/steroid-dependent chronic obstructive pulmonary disease)
14. Patients being taken up for liver transplant
15. Refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival | Day 21

SECONDARY OUTCOMES:
Improvement in cerebral edema and hepatic encephalopathy | Day 5
  Cerebral edema reduction will be assessed by a composite of clinical signs and bedside monitoring tools which includes
  1. Reduction in optic nerve sheath diameter below 4.5mm
  2. Improvement in EEG
  3. Reduction in hepatic encephalopathy to grade 2 or below
  4. Improvement in near-infrared spectroscopy by 20% from baseline or >45
  5. Reduction in ammonia by 25% at 24 hours
Improvement in cerebral edema and hepatic encephalopathy | Day 14
  Cerebral edema reduction will be assessed by a composite of clinical signs and bedside monitoring tools which includes
  1. Reduction in optic nerve sheath diameter below 4.5mm
  2. Improvement in EEG
  3. Reduction in hepatic encephalopathy to grade 2 or below
  4. Improvement in near-infrared spectroscopy by 20% from baseline or >45
  5. Reduction in ammonia by 25% at 24 hours
Duration of mechanical ventilation in both groups | 28 days
Duration of ICU stay in both groups | 28 days
Impact on arterial lactate | 6 hours
  Reduction or increase in arterial lactate by atleast 10% from baseline (at initiation of CRRT) would be recorded
Impact on arterial lactate | 12 hours
  Reduction or increase in arterial lactate by atleast 10% from baseline (at initiation of CRRT) would be recorded
Impact on arterial lactate | 24 hours
  Reduction or increase in arterial lactate by atleast 10% from baseline (at initiation of CRRT) would be recorded
Impact on arterial lactate | Day 5
  Reduction or increase in arterial lactate by atleast 10% from baseline (at initiation of CRRT) would be recorded
Impact on arterial lactate | Day 14
  Reduction or increase in arterial lactate by atleast 10% from baseline (at initiation of CRRT) would be recorded
Improvement in SIRS | Day 5
  Improvement in SIRS is defined reduction in SIRS by atleast one component or its resolution.
Effect on systemic hemodynamics | 24 hours
  Delta change in systemic hemodynamics ( as assessed by systemic vascular resistance) after intervention in both groups will be recorded.
Effect on systemic hemodynamics | Day 5
Effect on pulmonary function | 24 hours
  Pulmonary functions (assessed by measurement of extravascular lung water index and pulmonary vascular permeability index and PaO2/Fi02 ratio after intervention in both groups will be recorded.
Effect on pulmonary function | Day 5
  Pulmonary functions (assessed by measurement of extravascular lung water index and pulmonary vascular permeability index and PaO2/Fi02 ratio after intervention in both groups will be recorded.
Effect on endotoxin. | 5 days
  The delta change in endotoxin will be recorded.
Effect on DAMPS. | 5 days
  The delta change in DAMPS will be recorded.
Effect on pro-inflammatory cytokines. | 12 hours
  The delta change in pro-inflammatory cytokines will be recorded.
Effect on pro-inflammatory cytokines. | 5 days
  The delta change in pro-inflammatory cytokines will be recorded.
Effect on endothelial functions. | 5 days
  Effect on endothelial functions would be assessed by measurement of endothelin-1, angiopoietin-2, ADAMTs and von-willebrand factor
Effect on coagulation. | 5 days
  Effect on coagulation would be assessed by incidence of bleeding events, delta change in coagulation parameters as assessed by rotational thromboelastometry
To study the safety of therapy (incidence of intradialytic hypotension, impairment of coagulation, hypothermia) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided